CLINICAL TRIAL: NCT01500304
Title: Feasibility and Safety of Minimally Invasive Inguinal Lymph Node Dissection in Patients With Melanoma
Brief Title: Minimally Invasive Groin Dissection for Melanoma
Acronym: SAFE-MILND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James W. Jakub, Breast and Melanoma Surgery Section Head, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007790
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Melanoma
Keywords: Melanoma; Lymph Nodes; Lymph Node Dissection; Minimally invasive
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Minimally invasive surgery (Experimental): Minimally invasive inguinal lymph node dissection is a 10-step technique to provide novel inguinal lymph node staging and treatment.
  Interventions: Procedure: Minimally invasive inguinal lymph node dissection

INTERVENTIONS:
Procedure: Minimally invasive inguinal lymph node dissection — Operative intervention will be a minimally invasive inguinal lymphadenectomy, which is a three trocar technique to the inguinal dissection, that respects the same anatomic boundaries as the conventional open procedure
  Other Names: SAFE MILND

SUMMARY:
The purpose of this this study is to determine if a structured educational training program is successful in teaching surgeons a new operative technique. It will then be determined if this new operative technique is safe.

DETAILED DESCRIPTION:
This study is a multi-center, Phase 1 clinical trial to determine the safety and feasibility of minimally invasive inguinal lymph node dissection for patients with melanoma. Licensed surgeons who have undergone special training, including a course at the Mayo Clinic Rochester in minimally invasive lymph node dissection (MILND) will perform the new procedure at their home institutions. The study will characterize the learning curve of MILND in the clinical setting, and evaluate the safety of the new operative technique.

The hypotheses for this study are: 1) minimally invasive groin dissection is a safe procedure. 2) a structured educational training program is a feasible and effective method to train practicing surgeons in this novel procedure and 3) pre-course generic laparoscopic technical skills correlate with minimally invasive superficial groin dissection performance in a clinical setting, including operative oncologic standards and safety metrics.

ELIGIBILITY:
Inclusion criteria:

* Malignant melanoma present in an inguinal nodal basin requiring superficial inguinal lymph node dissection.
* Plan for superficial inguinal dissection alone or combined superficial inguinal and deep pelvic node dissection is acceptable.
* Clinical or radiographic evidence of superficial inguinal lymph node disease or a prior positive single lymph node biopsy of the superficial inguinal basin as an indication for superficial inguinal lymph node disease is acceptable.
* Patients must be Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 and be healthy enough to undergo a general anesthetic (no epidural or spinal anesthetics).
* Female patients of child bearing age must have a negative pregnancy test, be surgically sterile or post-menopausal greater than 1 year.
* Patients must be able to return to surgical facility for 30 and/or 90 day (+/- 20 days) for follow-up appointment.

Exclusion Criteria:

* Prior ipsilateral superficial inguinal lymph node dissection
* Invasion or ulceration of inguinal nodal disease into the overlying skin
* Prior radiation therapy to the same regional nodal basin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proficiency score per surgery | Approximately 90 days following surgical procedure
  The proficiency score is a function of the lymph nodes pathologically identified, the amount of blood transfused and the operative time. The range is 0 to 3, with higher proficiency in performing the procedure being 3.

SECONDARY OUTCOMES:
Morbidity and percentage of patients converted to open surgical procedure | Approximately 90 days following surgical procedure
  Perioperative morbidity will be prospectively collected and reported.Percentage of participants that require conversion from MILND to open procedure (standard of care). Conversion to the open procedure is required if the operation is not progressing, an adequate oncologic procedure cannot be completed or if bleeding is encountered that cannot be safety controlled videoscopically.

CONTACTS AND LOCATIONS:
Overall Officials: James Jakub, MD, Principal Investigator — Mayo Clinic
Locations (11):
- United States (11):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - John Wayne Cancer Institute, Santa Monica, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Background] Jakub JW, Reintgen DS, Shivers S, Pendas S. Regional node dissection for melanoma: techniques and indication. Surg Oncol Clin N Am. 2007 Jan;16(1):247-61. doi: 10.1016/j.soc.2006.10.012. PMID 17336247
- [Background] Abbott AM, Grotz TE, Rueth NM, Hernandez Irizarry RC, Tuttle TM, Jakub JW. Minimally invasive inguinal lymph node dissection (MILND) for melanoma: experience from two academic centers. Ann Surg Oncol. 2013 Jan;20(1):340-5. doi: 10.1245/s10434-012-2545-6. Epub 2012 Aug 9. PMID 22875645
- [Derived] Jakub JW, Terando AM, Sarnaik A, Ariyan CE, Faries MB, Zani S Jr, Neuman HB, Wasif N, Farma JM, Averbook BJ, Bilimoria KY, Grotz TE, Allred JB, Suman VJ, Brady MS, Tyler D, Wayne JD, Nelson H. Safety and Feasibility of Minimally Invasive Inguinal Lymph Node Dissection in Patients With Melanoma (SAFE-MILND): Report of a Prospective Multi-institutional Trial. Ann Surg. 2017 Jan;265(1):192-196. doi: 10.1097/SLA.0000000000001670. PMID 28009745
- [Derived] Jakub JW, Terando AM, Sarnaik A, Ariyan CE, Faries MB, Zani S Jr, Neuman HB, Wasif N, Farma JM, Averbook BJ, Bilimoria KY, Allred JB, Suman VJ, Grotz TE, Zendejas B, Wayne JD, Tyler DS. Training High-Volume Melanoma Surgeons to Perform a Novel Minimally Invasive Inguinal Lymphadenectomy: Report of a Prospective Multi-Institutional Trial. J Am Coll Surg. 2016 Mar;222(3):253-60. doi: 10.1016/j.jamcollsurg.2015.11.010. Epub 2015 Nov 25. PMID 26711792